CLINICAL TRIAL: NCT02423811
Title: To Study the Effect of Fursultiamine in Esophageal Squamous Cell Carcinoma Patients Who Receive Concurrent Chemoradiotherapy
Brief Title: Fursultiamine in Esophageal Squamous Cell Carcinoma Patients Who Receive Concurrent Chemoradiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-104-105
Record Dates: First submitted 2015-04-19; First posted 2015-04-22 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2015-04

CONDITIONS: Cancer Stem Cell
MeSH Terms: interventions — Fursultiamin

ARMS (1):
- CCRT plus Fursultiamine (Experimental): Fursultiamine 100mg tid, po Radiotherapy 36Gy/18Fx Chemotherapy will include Cisplatin and 5-FU. Cisplatin 60-75 mg/m2 on days 1 and 29 with standard prehydration and antiemetic therapy.
  5-FU 600-1000 mg/m2day administered as a continuous intravenous infusion for 96 hours after completion of the cisplatin on days 1 through 4 and 29 through 32
  Interventions: Dietary Supplement: Fursultiamine

INTERVENTIONS:
Dietary Supplement: Fursultiamine — Use of Fursultiamine in addition to CCRT

SUMMARY:
Esophageal cancer is a common and fatal malignancy. It is the eighth most common incident cancer and the sixth leading cause of cancer death in the world. In Taiwan, esophageal cancer was newly diagnosed in 2199 patients and was the cause of 1507 deaths in 2011. Squamous cell carcinoma is the predominant histological tumor type, accounting for about 90% of the cases. Esophageal squamous cell carcinoma (ESCC) is an aggressive disease, characterized with extensive local growth and frequent metastases. Concurrent chemoradiotherapy (CCRT) with or without surgery is the treatment option for locally advanced ESCC. Further, target therapy is used in conjunction with CCRT and surgery in ESCC since several years ago. However, the therapeutic outcomes are not satisfactory due to the emergence of chemo-radioresistance. It is imperative to investigate new biomarkers and to find novel treatment targets in ESCC.

A small population of tumor-initiating cells or cancer stem cells (CSCs) possess some biological functions like normal stem cells, including self-renewal, asymmetric cell division, slowly proliferation rate and drug-resistance. CSCs from many primary tumors and cell lines express specific stem cell markers, including Oct4, Sox2, Nanog, CD133 (promimin-1), Nestin, CD44 ,CD24, ALDH (Aldehyde dehydrogenase) and c-Kit. There are many evidences that CSCs are responsible for tumor initiation, progression and metastasis. CSCs are also believed to have important roles in cancer recurrence due to their resistance to anti-cancer drugs and radiation. CSCs express high levels of ATP-binding cassette (ABC) transporters. ABC transporter can pump cytotoxic drugs out of cells and is one important mechanism of multidrug resistance in CSCs. In addition, CSCs have high reactive oxygen species (ROS) scavenger expression to remove ROS produced from irradiation therapy.

Fursultiamine (also known as thiamine tetrahydrofurfuryl disulfide, TTFD) is a derivative of vitamin B and currently used for nutrition supplement. The investigators have identified that Fursultiamine suppressed OCT-4, SOX-2, NANOG expression and decreased ABCB1 and ABCG2 in tumor sphere of ESCC cell lines. In this project, the investigators will conduct a prospective phase II study to investigate the effect of Fursultiamine combined with CCRT in ESCC patients. Stem cell markers in clinical specimens collected before and after CCRT will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed stage II and III esophageal squamous cell carcinoma

Exclusion Criteria:

* ECOG≧2;
* impaired function of lung, liver, kidney or bone marrow

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Forn-Chia Lin, M.D., Ph.D., Principal Investigator — Department of Radiation Oncology, National Cheng Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan